CLINICAL TRIAL: NCT00344617
Title: Off-Label Use of AVASTIN (BEVACIZUMAB)Intravitreal Injection For the Treatment of Serosanguinous Maculopathy
Brief Title: Off-Label AVASTIN (BEVACIZUMAB) For Serosanguinous Maculopathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore National Eye Centre (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R452/01/2006
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Choroidal Neovascularisation; Polypoidal Choroidal Vasculopathy
Keywords: Choroidal neovascularisation; Polypoidal choroidal vasculopathy; Intravitreal injection; Avastin
MeSH Terms: conditions — Choroidal Neovascularization; Polypoidal Choroidal Vasculopathy | interventions — Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab (tradename: Avastin)

SUMMARY:
To assess the use of Avastin for the management of serosanguinous maculopathy

DETAILED DESCRIPTION:
METHODOLOGY

Patients will be recruited from the vitreoretinal clinics at SNEC. After initial assessment, clinically and angiographically, the patient will be counselled with regards to diagnosis, prognosis and management options, including the option of intravitreal Avastin.

Inclusion criteria:

1. All subfoveal/juxtafoveal CNV and PCV (polypoidal choroidal vasculopathy) who are not eligible for other treatment options (compassionate use)
2. CNV and PCV lesions which have failed PDT, conventional argon laser photocoagulation (salvage use)
3. CNV and PCV lesions treatable with PDT, but cannot afford or refused

Exclusion criteria:

1. Patients with uncontrolled hypertension (systolic BP greater than 150mmHg or diastolic BP greater than 90mmHg
2. History of thrombolic events such as myocardial infarction or cerebral vascular accident
3. Renal abnormalities as defined by established history of chronic renal disease or renal failure as well as patients requiring dialysis
4. Recent (as defined as the past 28 days) or planned (as defined as the next 3 months) surgery.
5. Coagulation abnormalities, including anti-coagulant medication other than aspirin
6. Patients with peptic ulcer disease
7. Pregnant or lactating females

If the patient is agreeable to the intravitreal treatment protocol, he/she will be assessed systemically for fitness for the therapy. The serosanguinous maculopathy will be subtyped by angiographic findings to predominantly classic (>50% classic component) lesions, minimally classic (<50% classic component) lesions, occult lesions and polypoidal choroidal vasculopathy (PCV).

If the patient is eligible for the intravitreal treatment protocol, he/she will receive 1mg of Avastin intravitreally. This will be performed under aseptic technique. (See attached 'Intravitreal Injection Protocol'). The injections will be repeated every 8-10 weeks for a total of 3 treatments.

END OF TREATMENT

If the central retinal thickness is reduced by >50%, or if there is imrpovement/stablisiation of vision, or if an adverse effect (such as elevation of BP) is encountered, the treating physician can elect to withhold the Avastin treatment.

On review at the 8 and 16 weeks, the physician can elect to perform additional intravitreal Avastin treatment if any of the following should arise

1. Loss of VA of at least 5 letters at 2 sequential visits within 2 weeks, which is associated with increased leakage from the CNV seen on angiography or OCT
2. Increase in OCT central retinal thickness by >100um
3. Onset of a new macular haemorrhage
4. Development of a new classic CNV membrane
5. Ocular outcome measurements
6. Change from baseline in VA, i.e. gain or loss of 5 letters (1 line), 15 letters (3 lines) or 30 letters (6 lines)

Secondary outcomes

1. Change in OCT measured central retinal thickness
2. Correlation in change in central retinal thickness and change in VA

Once informed consent has been obtained for intravitreal Avastin therapy, the patient will be assessed for the fitness to indergo the treatment. Baseline systemic & ocular assessments will be performed. Systemic assessment will include blood pressure measurement, electrocardiogram (ECG) and blood investigations (full blood count, prothrombin time, partial thromboplastin time, bleeding time)

Once deemed fit, the patient will receive Injection 1 of intravitreal Avastin (Refer Intravitreal Injection Protocol)

The patient will then be reviewed at 1 week post-injection and then monthly for the first 2 months. Investigations at these visits will include logMAR BCVA, biomicroscopy, FFA and OCT.

At the time point of 8-10 weeks, the patient will undergo Injection 2. Followed by review at 1 week post-injection and monthly for 2 months with the same investigations as stated above.

At 16-20 weeks, the patient will receive the last treatment, Injection 3, with similar post-injection visits and investigations.

If the central retinal thickness is reduced by >50%, or if there is imrpovement/stablisiation of vision, or if an adverse effect (such as elevation of BP) is encountered, the treating physician can elect to withhold the second and/or third Avastin treatment. Hence, each patient will receive at least 1 injection of Avastin and up to a maximum of 3 injections.

ELIGIBILITY:
Inclusion Criteria:

1. All subfoveal/juxtafoveal CNV and PCV (polypoidal choroidal vasculopathy) who are not eligible for other treatment options (compassionate use)
2. CNV and PCV lesions which have failed PDT, conventional argon laser photocoagulation (salvage use)
3. CNV and PCV lesions treatable with PDT, but cannot afford or refused

Exclusion Criteria:

1. Patients with uncontrolled hypertension (systolic BP greater than 150mmHg or diastolic BP greater than 90mmHg
2. History of thrombolic events such as myocardial infarction or cerebral vascular accident
3. Renal abnormalities (as defined by established history of chronic renal disease or renal failure as well as patients requiring dialysis).
4. Recent (as defined as the past 28 days) or planned (as defined as the next 3 months) surgery.
5. Coagulation abnormalities, including anti-coagulant medication other than aspirin
6. Patients with peptic ulcer disease
7. Pregnant or lactating females

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-06; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in VA, i.e. gain or loss of 5 letters (1 line), 15 letters (3 lines) or 30 letters (6 lines)

SECONDARY OUTCOMES:
Change in OCT measured central retinal thickness
Correlation in change in central retinal thickness and change in VA

CONTACTS AND LOCATIONS:
Overall Officials: Chong-Lye Ang, FRCOphth, Principal Investigator — Singapore National Eye Centre

REFERENCES:
- [Background] Michels S, Rosenfeld PJ, Puliafito CA, Marcus EN, Venkatraman AS. Systemic bevacizumab (Avastin) therapy for neovascular age-related macular degeneration twelve-week results of an uncontrolled open-label clinical study. Ophthalmology. 2005 Jun;112(6):1035-47. doi: 10.1016/j.ophtha.2005.02.007. PMID 15936441
- [Background] Rosenfeld PJ, Moshfeghi AA, Puliafito CA. Optical coherence tomography findings after an intravitreal injection of bevacizumab (avastin) for neovascular age-related macular degeneration. Ophthalmic Surg Lasers Imaging. 2005 Jul-Aug;36(4):331-5. PMID 16156152